CLINICAL TRIAL: NCT04186377
Title: A Study of the Effectiveness of Local S26E Extract Application for Diabetic Foot Ulcer Healing
Brief Title: Application of S26E for Diabetic Foot Ulcer Healing
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to recruit subjects
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Alexandros Kokkinos, Associate Professor in Internal Medicine, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S26E for neuropathic ulcers
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Diabetic Foot; Neuropathic Foot Ulcer; Chronic Diabetic Ulcer of Left Foot (Diagnosis); Chronic Diabetic Foot Ulcer of Right Foot
MeSH Terms: conditions — Diabetic Foot; Disease | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-of-care managed group (Active Comparator): This group will receive the optimal standard-of-care for neuropathic/neuroischemic diabetic foot ulcers
  Interventions: Other: Standard-of-care for neuropathic/neuroischemic diabetic foot ulcers
- S26E (Experimental): This group will receive the optimal standard-of-care for neuropathic/neuroischemic diabetic foot ulcers plus daily S26E application
  Interventions: Other: Standard-of-care for neuropathic/neuroischemic diabetic foot ulcers; Drug: S26E

INTERVENTIONS:
Other: Standard-of-care for neuropathic/neuroischemic diabetic foot ulcers — Optimization of glycemic control, off-loading, local debridement as needed, atraumatic surface scrubbing, saline washing and sterile dressing
Drug: S26E — Daily application of S26E extract on wound site
  Arms: S26E

SUMMARY:
A randomized, controlled open-label, parallel group study to examine the effectiveness of a local application of the kalahari melon (Citrullus lanatus) seed oil for the healing of non-infected diabetic foot ulcers.

DETAILED DESCRIPTION:
This is a randomized, controlled open-label, parallel group study of 12 weeks duration aimed to examine the effectiveness of a local application of the kalahari melon (Citrullus lanatus) seed oil (S26E) for the healing of non-infected chronic (>12 weeks) diabetic foot ulcers. The S26E is a natural extract rich in unsaturated (such as linoleic, oleic, palmitic and static) fatty acids which have shown promise in the promotion of wound healing by modulating the migration and functional properties of inflammatory cells in wound cites as well as the production of inflammatory cytokines. The safety of topical S26E application on human skin has been clinically demonstrated.

Eligible participants will be adults patients with diabetes mellitus (DM) type 1 or 2 and chronic (persistent for >12 weeks after initial presentation) neuropathic or neuroischaemic non-infected diabetic foot ulcers. Following recruitment and randomization (on a 1:1 ratio) eligible patients will attend the study site on weekly intervals. After a run-in period of 2 weeks (visits 1-2) during which all participants will receive the optimal standard-of-care for neuropathic/neuroischaemic diabetic ulcers (incl. optimization of glycemic control, off-loading, local debridement as needed, atraumatic surface scrubbing, saline washing and sterile dressing) eligibility will be reassessed. Participants who will continue in the study will receive standard of care (control group) or standard of care plus daily local S26E application on ulcer (intervention group) (visits 3-12). After visit 12 the application of S26E will be terminated and all participants will receive an additional follow up visit 4 weeks later (final visit). Efficacy end-points will be assessed at the end of the of 12 weeks of observation (Visit 12)

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 Diabetes Mellitus
* Body Mass Index <40 kg/m2
* Glycated Hemoglobin (HbA1c) <10%
* Presence of a diabetic foot ulcer with the following features i) Owing to chronic peripheral sensorimotor diabetic neuropathy, with or without peripheral arterial disease (critical ischemia excluded as indexed by an Ankle-Brachial index <0.4 ) ii) Persistence for >12 weeks iii) Already following an adequate off-loading method

Exclusion Criteria:

* Presence of clinical signs of infection
* Inability or refusal to follow off-loading methods
* Ulcer surface area decline by >15% during the run-in period
* Malignant disease (non-melanoma skin malignancy and healed thyroid malignancies excluded)
* Acute Charcot arthropathy
* Serious chronic Hepatic (Child-Pugh B or C), Renal (stage 4-5 CKD) or Heart (NYHA 3-4) disease
* Known hypersensitivity to the product or its contents
* Any random glucose measurement >350 mg/dl during the run-in period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Change of ulcer surface area | 12 weeks after enrollment in the study
  % change of ulcer surface area

SECONDARY OUTCOMES:
Percentage of completely healed ulcers | 12 weeks after enrollment in the study
  Percentage of participants to achieve ulcer healing within the observation period
Incidence of adverse events | 12 weeks after enrollment in the study
  Incidence of product-related adverse events (local or systemic infection, local hypersensitivity reactions)
Incidence of amputations | 12 weeks after enrollment in the study
  Number of patients that required an amputation

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes Clinical Research Laboratory, 1st Department of Propaedeutic Internal Medicine, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheikhyoussef N, Kandawa-Schulz M, Bock R, de Koning C, Cheikhyoussef A, Hussein AA. Characterization of Acanthosicyos horridus and Citrullus lanatus seed oils: two melon seed oils from Namibia used in food and cosmetics applications. 3 Biotech. 2017 Oct;7(5):297. doi: 10.1007/s13205-017-0922-3. Epub 2017 Aug 31. PMID 28868224
- [Background] Silva JR, Burger B, Kuhl CMC, Candreva T, Dos Anjos MBP, Rodrigues HG. Wound Healing and Omega-6 Fatty Acids: From Inflammation to Repair. Mediators Inflamm. 2018 Apr 12;2018:2503950. doi: 10.1155/2018/2503950. eCollection 2018. PMID 29849484
- See also: Related Info — https://www.researchgate.net/publication/224864433_Oil_and_Fatty_Acid_Contents_in_Seed_of_Citrullus_lanatus_Schrad